CLINICAL TRIAL: NCT00370383
Title: A Phase 2 Study Comparing Sequential Satraplatin and Erlotinib to Single-Agent Erlotinib in Patients ≥ 70 Years of Age With Unresectable Stage 3 OR 4 Non-Small Cell Lung Cancer as 1st-Line Therapy
Brief Title: A Study Comparing Sequential Satraplatin & Erlotinib to Erlotinib in Unresectable Stage 3/4 Non-small-cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAT2-05-07
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: Non Small Cell Lung Cancer; PATIENTS ≥ 70 YEARS WITH UNRESECTABLE STAGE 3 OR 4 NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; satraplatin

ARMS (2):
- Satraplatin (Experimental): Satraplatin administered orally once daily for 5 consecutive days followed by erlotinib for 14 consecutive days
  Interventions: Drug: Erlotinib; Drug: Satraplatin
- Erlotinib (Experimental): Erlotinib administered orally once daily. Erlotinib - [6,7-Bis(2-methoxy-ethoxy)-quinazolin-4-y]- (3-ethynyl-phenyl)amine hydrochloride, molecular weight 393.4. This is a small molecule that competes with the binding of ATP to the intracellular tyrosine kinase domain of EGFR, thereby inhibiting receptor autophosphorylation and blocking downstream signal transduction.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — erlotinib 150 mg/day once daily
Drug: Satraplatin — satraplatin 100 mg/m2 orally once daily for 5 consecutive days (days 1-5)followed by erlotinib 150mg/day for 14 consecutive days (days 8-21).
  Satraplatin JM-216, bis-aceto-ammine dischlorocyclohexylamine platinum)is a third-generation platinum analogue with activity following oral administration. The molecular formula for satraplatin is C10H22N2Cl2O4Pt, which is structured as an octahedral platinum compound.
  Arms: Satraplatin

SUMMARY:
Patients ≥ 70 years of age with locally advanced unresectable or metastatic non-small cell lung cancer (NSCLC) frequently do not receive systemic cytotoxic chemotherapy due to concerns regarding their inability to tolerate treatment. Epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKIs) are agents with favorable toxicity profiles that have shown activity in patients with NSCLC. Erlotinib as a single-agent is currently approved for the treatment of patients with NSCLC whose disease has progressed following one prior course of chemotherapy and is currently being evaluated in NSCLC patients who have not received prior systemic treatment. However, when studied with combination chemotherapy in the first-line setting, continuous daily administration of erlotinib did not result in improved patient survival. Further clinical and in vitro data suggest that the sequencing of cytotoxic chemotherapy with EGFR TKIs is important to maximize their therapeutic potential when administered in combination.

Satraplatin is an oral, investigational anticancer drug that is a member of the platinum-based class of chemotherapy drugs. Platinum-based drugs have been clinically proven to be one of the most effective classes of anticancer therapies. Unlike the currently marketed platinum-based drugs, satraplatin can be given orally and is currently being evaluated in a pivotal phase 3 clinical trial as 2nd-line therapy for patients with hormone refractory prostate cancer.

The rationale for this study is to develop an active and well-tolerated oral regimen for patients ≥ 70 years of age with NSCLC. Administration of the study drugs will be sequenced with satraplatin administered on days 1-5 and erlotinib on days 8-21 of each 28-day cycle. The primary endpoint will be progression-free survival (PFS). Patients will be randomized to treatment with either the experimental regimen or single-agent continuous erlotinib.

DETAILED DESCRIPTION:
Erlotinib as a single-agent is currently approved for the treatment of patients with NSCLC whose disease has progressed following one prior course of chemotherapy and is currently being evaluated in NSCLC patients who have not received prior systemic treatment. However, when studied with combination chemotherapy in the first-line setting, continuous daily administration of erlotinib did not result in improved patient survival. Further clinical and in vitro data suggest that the sequencing of cytotoxic chemotherapy with EGFR TKIs is important to maximize their therapeutic potential when administered in combination.

Satraplatin is an orally administered platinum analogue that has shown promising single-agent activity in multiple tumor types including prostate, ovarian, and small cell lung cancer. Additionally, the single-agent activity of satraplatin in NSCLC is similar to that of other commonly used platinum agents used to treat NSCLC. However, satraplatin is better tolerated than cisplatin, causing less renal toxicity and ototoxicity, and it can be administered in the outpatient setting. From a toxicity profile, it is more similar to carboplatin in that myelosuppression is its dose limiting toxicity (DLT). Satraplatin is currently being evaluated in a pivotal phase 3 clinical trial as 2nd-line therapy for patients with hormone refractory prostate cancer.

The rationale for this study is to develop an active and well-tolerated oral regimen for patients ≥ 70 years of age with NSCLC who may not be candidates for aggressive combination systemic chemotherapy. Administration of the study drugs will be sequenced with satraplatin administered on days 1-5 and erlotinib on days 8-21 of each 28-day cycle. As erlotinib has shown an advantage in survival without a commensurate improvement in response rate, the primary endpoint will be progression-free survival (PFS); thus patients will be randomized to treatment with either the experimental regimen or single-agent continuous erlotinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC (squamous cell carcinoma, adenocarcinoma, or large cell carcinoma). Cytologic specimens obtained by brushings, washings or needle biopsy with aspiration are acceptable. Mixed tumors with small cell anaplastic elements are not eligible.
* Patients who have unresectable stage III or stage IV disease are eligible. Patients with stage III disease should be ineligible for combined modality therapy (i.e. pleural effusions, pericardial effusions, etc.). Patients with earlier stage NSCLC that has recurred after prior surgery are eligible.
* Age ≥ 70 years old.
* ECOG performance status 0-1
* Prior treatment with systemic therapy is allowed provided the following criteria are met:

  * No EGFR targeted therapy (TKI or antibody)
  * No prior platinum agent.
  * Neoadjuvant, adjuvant, or part of a combined modality regimen (i.e., not for metastatic disease)
  * Completion > 6 months prior to enrollment onto this study.
  * Patients who have had previous radiation therapy (RT) as definitive therapy for locally NSCLC are eligible only if the following criteria are met:
  * Site of tumor recurrence is outside of the original RT port unless there is incontrovertible evidence of disease progression within the portal
  * All side effects from RT must have resolved prior to enrollment.
  * Completion of RT ≥ 4 weeks prior to enrollment.
  * Previous radiation must have treated < 30% of active bone marrow.
  * Patients who have undergone thoracotomy must have fully recovered from surgery and cannot start treatment until at least three weeks after their operative procedure.
* Adequate hematological function as noted by:

  * Absolute neutrophil count (ANC) > 1,500/ L
  * Platelets > 100,000/ L
  * Hemoglobin > 10 g/dl. Patients may be transfused or receive erythropoietin to maintain or exceed this level.
* Adequate hepatic and renal function as noted by:

  * Bilirubin < 1.5 x ULN
  * Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) < 2.5 x ULN.
  * Serum creatinine ≤ 1.5mg/dL or calculated (or measured) glomerular filtration rate ≥ (GFR)50 ml/min.
  * Patients with both measurable and non-measurable disease (as per Response Criteria in Solid Tumors (RECIST)) may be enrolled.

Exclusion Criteria:

* Concurrent invasive malignancy requiring ongoing therapy.
* Metastatic brain or meningeal tumors, unless the patient is > 1 month from definitive therapy, is clinically stable with respect to the tumor at the time of study entry, is not receiving steroid therapy or taper, and is not receiving anti-convulsant medications (that were started for the brain metastases).
* Previous treatment with either platinum-based chemotherapy agents or prior EGFR targeting agents.
* Peripheral neuropathy > grade 1.
* Hearing loss or tinnitus > grade 2
* Obstructive pulmonary disease or symptoms > grade 3.
* A history of cardiac disease as defined by malignant hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous six months, or symptomatic uncontrolled cardiac arrhythmias.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-07; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To compare Progression-Free Survival (PFS) in patients ≥ 70 years of age, PS 0-1, with advanced or metastatic NSCLC in patients treated with a first-line regimen of either sequential satraplatin and erlotinib or continuous single-agent erlotinib. | January, 2008

SECONDARY OUTCOMES:
To assess Overall Survival in patients ≥ 70 years of age, PS 0-1, with advanced or metastatic NSCLC in patients treated with a first-line regimen of either sequential satraplatin and erlotinib or continuous single-agent erlotinib. | January, 2008
To compare response rates. | January, 2008
To compare the toxicity profiles between patients treated with satraplatin and erlotinib and single-agent erlotinib | January, 2008

CONTACTS AND LOCATIONS:
Overall Officials: Corey Langer, MD, Principal Investigator — Fox Chase Cancer Center
Locations (16):
- United States (11):
  - Pacific Cancer Medical Center, Anaheim, California
  - Scripps Clinic, La Jolla, California
  - Kenmar Research Institute, Los Angeles, California
  - Memorial Cancer Institute, Hollywood, Florida
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Highlands Oncology Group, Bentonville, Ohio
  - Gabrail Cancer Center, Canton, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Signal Point Hematology/Oncology, Middleton, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Canada (2):
  - McGill University, Montreal
  - Princess Margaret Hospital, Toronto
- Chile (3):
  - Hospital San Borja Arriaran, Santiago
  - Instituto Nacional del Cancer, Santiago
  - Research Center, Santiago